CLINICAL TRIAL: NCT03481959
Title: Effectiveness of Methylphenidate Late Formula to Reduce Cannabis Use in Young Cannabis-Related Patients and Attention Deficit Disorder Hyperactivity
Acronym: METHACAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recrutement in the study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P140313
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2020-11

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: TDAH; Methylphenidate; Cannabis
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Marijuana Abuse | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylphenidate (Experimental): Methylphenidate delay shape, 10 and 30 mg capsules. Treatment should be started at a dose of 10 mg per day or 20 mg/d (depending on the weight of patients), with increasing weekly, according to the clinical tolerance, in order to get an effective dose on the symptoms of ADHD to S4, not more than 1 mg/kg/d (capped at 60 mg/d).
  Interventions: Drug: Methylphenidate
- Matching Placebo (Placebo Comparator)
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate delay shape, 10 and 30 mg and matching Placebo capsules. Treatment should be started at a dose of 10 mg per day or 20 mg/d (depending on the weight of patients), with increasing weekly, according to the clinical tolerance, in order to get an effective dose on the symptoms of ADHD to S4, not more than 1 mg/kg/d (capped at 60 mg/d).
  This gradual dose treatment will be resumed in the same manner in M3 at the beginning of the phase in open, allowing the respect of the average of the ADHD support (no), without loss of chance for the Group at 3 months, because it is customary to discontinue treatment during holiday periods).
  Arms: Methylphenidate
Other: Matching Placebo — Methylphenidate delay shape, 10 and 30 mg and matching Placebo capsules. Treatment should be started at a dose of 10 mg per day or 20 mg/d (depending on the weight of patients), with increasing weekly, according to the clinical tolerance, in order to get an effective dose on the symptoms of ADHD to S4, not more than 1 mg/kg/d (capped at 60 mg/d).
  This gradual dose treatment will be resumed in the same manner in M3 at the beginning of the phase in open, allowing the respect of the average of the ADHD support (no), without loss of chance for the Group at 3 months, because it is customary to discontinue treatment during holiday periods).
  Arms: Matching Placebo

SUMMARY:
Abuse of psychoactive substances is a behavior belonging to the field of risk behaviors that begins and takes place during adolescence. These risk behaviors are a major public health problem in France and worldwide.

Cannabis is the first illicit drug consumed by adolescents in France. His experimentation progresses rapidly between 11 and 17 years. The relationship between cannabis use and mental health has been shown by several studies. In particular Attention Deficit Hyperactivity Disorder (ADHD), characterized by attention deficit, impulsivity and disabling motor hyperactivity and beginning before 12 years of age (DSM-5), is a major risk factor for the consumption of cannabis. ADHD is a common condition (9% of children and 5% of adults), but often undiagnosed or untreated. It has been shown that the treatment of ADHD in childhood protects the consumption of psychoactive products during adolescence or adulthood. However, to our knowledge there is no study showing that treatment with methylphenidate in an ADHD patient - not treated - but already a cannabis user, was a positive prognostic factor in the decrease in cannabis use.

DETAILED DESCRIPTION:
Abuse of psychoactive substances is a behavior belonging to the field of risk behaviors that begins and takes place during adolescence. These risk behaviors are a major public health problem in France and worldwide.

Cannabis is the first illicit drug consumed by adolescents in France. His experimentation progresses rapidly between 11 and 17 years. The relationship between cannabis use and mental health has been shown by several studies. In particular Attention Deficit Hyperactivity Disorder (ADHD), characterized by attention deficit, impulsivity and disabling motor hyperactivity and beginning before 12 years of age (DSM-5), is a major risk factor for the consumption of cannabis. ADHD is a common condition (9% of children and 5% of adults), but often undiagnosed or untreated. It has been shown that the treatment of ADHD in childhood protects against the use of cannabis during adolescence or adulthood. However, there is no study showing that treatment with methylphenidate in an ADHD patient - not treated - but already a cannabis user, was a positive prognostic factor in the decrease in cannabis use.

Hypothesis: The hypothesis of this study is that patients diagnosed with ADHD and cannabis-treated patients treated with methylphenidate will decrease their number of days of cannabis use compared to ADHD patients receiving placebo.

Originality and Innovative There is no study showing that treatment with methylphenidate in an ADHD patient - not treated - but already a problematic cannabis user, was a positive prognostic factor in decreasing cannabis use.

Moreover, there is not enough team in addiction trained in the detection of attention deficit disorder which is now recognized as a factor of vulnerability for the development of addictions. This project is the opportunity for a training in the detection of the ADHD in the adolescent and the young adult of the professionals of the addiction and the setting up of a treatment by Methylphenidate as well as its handling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 and ≤ 25 years;
* Patients from 25 to 120 kg
* ADHD diagnosed according to the criteria of the DSM - V
* ADHD-RS-IV ≥ 28 test score;
* Without medication by methylphenidate for at least 6 months;
* Lack of psychiatries co-morbidities associated with a contraindication to treatment with methylphenidate (confirmed by MINI or MINI Kid); absence of BPD (tracked by the self-administered questionnaire MSI - BPD).
* Cannabis dependence objectified by a positive qualitative urinary dosage and a score ≥ 7 to CAST questionnaire;
* Consent of parents (child/teenager < 18 years) or young age if ≥ 18 years - patients of childbearing age agreeing to use a contraceptive method during the duration of the test

Exclusion Criteria:

Patients placed in child welfare (ASE).

* Pregnant patients or nursing
* No affiliation to a scheme of social security (beneficiary or beneficiary)
* Contraindications to treatment with methylphenidate :known hypersensitivity to methylphenidate or any of the excipients, glaucoma, pheochromocytoma,treatment by non selective irreversible inhibitors of the mono-amine oxidase (MAOI) and also for at least 14 days after stopping treatment with an MAOI because of the risk of hypertensive thrust,Treatment by other sympathomimetic indirect or sympathomimetic (oral and/or nasal way) alpha,Hyperthyroidism or wrong,diagnosis or history of severe depression, anorexia nervosa or disorders anorexia, suicidal tendencies, mood disorders, psychotic symptoms, mania, schizophrenia, psychopathic personality disorder, or limit (borderline), occlusal,diagnosis or history (affective) bipolar disorder severe (for type 1) and episodic (and poorly controlled), pre-existing cardiovascular disorders including severe hypertension, heart failure, pad angina, congenital heart disease with hemodynamic impact; cardiomyopathy, myocardial infarction, arrhythmias and channelopathies (disorders caused by a dysfunction of ion channels) that can potentially be life-threatening, pre-existence of disorders, stroke, cerebral aneurysm, vascular abnormalities, including stroke or Vasculitis and major Patient protected by law.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Number of days of use of cannabis | 12 weeks
  Number of days of use of cannabis in the past 21 days measured in 12 weeks by the TimeLine Follow Back (TLFB 21)

SECONDARY OUTCOMES:
Number of days of use of cannabis | 4,8,12 weeks and 12 months
  The average amount of daily consumption of cannabis within the past 21 days will be assessed from the TLFB 21-4, 8, 12 weeks and 12 months
Average daily consumption of cannabis in the last 21 days | 4,8,12 weeks and 12 months
  will be evaluated from the TLFB 21. The TLFB 21 makes it possible to quantify the number of daily cannabis
ADHD Rating scale IV score | 4,8,12 weeks and 12 months
  The scale evaluates the frequency of behavior, the level of behavioral discomfort and the developmental level.
advanced CAST score | one day, 12 weeks and one year
  The CAST is a 6-item scale, each of which describes use behaviors or problems encountered in the context of cannabis use
the score of the Hooked on nicotine checklist (HONC) | one day, 4,8,12 weeks and 12 months
  HONC is a self-administered questionnaire that assesses nicotine addiction.
the score of French version of the Tobacco Craving Questionnaire (FTCQ-12) | one day, 4,8,12 weeks and 12 months
  Evaluation of tobacco craving from the four primary factors of tobacco craving: emotionality, craving in anticipation of withdrawal relief or negative mood; waiting, compulsion and anticipation
Psychiatric comorbidities | one day, 12 weeks and 12 months
Consumption of other drugs | one day, 12 weeks and 12 months
Score of Overall Clinical Improvement Scale (CGI-S) | one day, 4,8,12 weeks and 12 months
  Measurement of symptom severity, response to treatment and efficacy of treatment in treatment studies of patients with mental disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Peyret Emmanuelle, PHD, Principal Investigator — APHP
Locations (1):
- Peyret, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boesen K, Paludan-Muller AS, Gotzsche PC, Jorgensen KJ. Extended-release methylphenidate for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2022 Feb 24;2(2):CD012857. doi: 10.1002/14651858.CD012857.pub2. PMID 35201607